CLINICAL TRIAL: NCT00896064
Title: A Study to Evaluate Safety and Immunogenicity of a Booster Dose of Two Formulations of GSK Biologicals' Pneumococcal Candidate Vaccine in Healthy Young Adults
Brief Title: Evaluation of a Booster Dose of Pneumococcal Vaccine Formulations in Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112993
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2017-04

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine; Streptococcus pneumoniae; Young adults
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Formulation 1 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A (formulation 1)
- Formulation 2 (Experimental)
  Interventions: Biological: Pneumococcal vaccine GSK2189242A (formulation 2)

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK2189242A (formulation 1) — One dose will be administered intramuscularly at Study Day 0.
  Arms: Formulation 1
Biological: Pneumococcal vaccine GSK2189242A (formulation 2) — One dose will be administered intramuscularly at Study Day 0.
  Arms: Formulation 2

SUMMARY:
The purpose of this study is to evaluate the safety, reactogenicity and immunogenicity of a booster dose of pneumococcal vaccines (GSK 2189242A) in young adults.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT 00707798)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 18 and 41 years old at the time of vaccination.
* Subjects who previously participated in the study NCT00707798 and received one of the two investigational GSK2189242A vaccine formulations during the primary study.
* Written informed consent obtained from the subject.
* Free of obvious health problems as established by medical history, clinical examination and clinical laboratory assessment before entering into the study.
* Female subjects of non-childbearing potential (defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause) may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after vaccination.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the vaccination, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting 30 days prior to the vaccination and ending one month (minimum 30 days) after vaccination.
* Administration of any pneumococcal vaccine other than the study vaccine during the period between end of study NCT00707798 and study vaccination.
* Bacterial pneumonia within the period between end of study NCT00707798 and study vaccination.
* Invasive pneumococcal disease (IPD) within the period between end of study NCT00707798 and study vaccination.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection (no laboratory testing required).
* History of thrombocytopenia or bleeding disorder.
* Anaphylactic reaction following the previous administration of the vaccine or history of reactions or allergic disease likely to be exacerbated by any component of the vaccine.
* Current serious neurologic or mental disorders.
* Inflammatory processes such as known chronic active infections (e.g. Hepatitis B, C).
* All past or current malignancies (excluding non-melanic skin cancer) and lymphoproliferative disorders.
* Acute disease at the time of enrolment/vaccination.
* Fever at the time of vaccination. Fever is defined as temperature >= 37.5°C on oral setting.
* Physical examination positive for acrocyanosis, jaundice, splenomegaly.
* Acute or chronic, clinically significant anaemia, pulmonary, cardiovascular, hematologic, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests, at the discretion of the investigator
* Administration of immunoglobulins and/or any blood products within the three months preceding vaccination or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.

Ages: 18 Years to 41 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-05-18; Primary Completion 2009-08-05 (Actual); Study Completion 2009-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 112993 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112993 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112993 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112993 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112993 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK2189242A Formulation 1 Group: Healthy male and female subjects, aged between 18 and 41 years old, who were previously primed with the GSK2189242A Formulation 1 vaccine during the 111651 study, received a booster dose of the GSK2189242A Formulation 1 vaccine, administered via intramuscular injection into the deltoid of the non-dominant arm, at Day 0.
- GSK2189242A Formulation 2 Group: Healthy male and female subjects, aged between 18 and 41 years old, who were previously primed with the GSK2189242A Formulation 2 vaccine during the 111651 study, received a booster dose of the GSK2189242A Formulation 2 vaccine, administered via intramuscular injection into the deltoid of the non-dominant arm, at Day 0.
Period: Overall Study
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Started | 22 | 21
Completed | 22 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.7 (4.80) | 23.9 (4.11) | 25.33 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 7 | 9 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White-Caucasian/European heritage | 22 | 21 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Grade 3 pain = significant pain at rest, pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 50 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Grade 3 Pain | 0 | 1
  Grade 3 Redness | 0 | 1
  Grade 3 Swelling | 1 | 0

2. Primary Outcome: Number of Subjects With Grade 3 and Vaccine-related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache, malaise, myalgia and fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = general symptom assessed by the investigator to be casually related to the study vaccination.
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 3 | 13
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 3 | 0
  Grade 3 Headache | 0 | 0
  Related Headache | 5 | 8
  Grade 3 Malaise | 0 | 0
  Related Malaise | 2 | 3
  Grade 3 Myalgia | 0 | 0
  Related Myalgia | 3 | 3
  Grade 3 Fever | 0 | 0
  Related Fever | 1 | 0

3. Primary Outcome: Number of Subjects With Grade 3 and Vaccine-related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Grade 3 AE(s) | 1 | 1
  Related AE(s) | 1 | 1

4. Primary Outcome: Number of Subjects With Any Vaccine-related Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Day 0 to Day 30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

5. Primary Outcome: Number of Subjects With Grade 3 Haematological or Biochemical Abnormalities
Description: Among haematological or biochemical abnormalities assessed were: Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Cholesterol, Creatine Phosphokinase (CRP), Hemoglobin decrease, Haemoglobin, Lactate dehydrogenase (LDH), Neutrophils, Red blood cells (RBC), Reticulocytes, White blood cells (WBC) and Overall parameters.
  Assessment of intensity: Grading of the haematological and biochemical parameters was performed using the standard Food and Drug Administration (FDA) Toxicity Grading Scale. Changes compared to normal reference ranges were graded: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening
Time Frame: At Days 1 and 6 post-booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  ALT, Day 1: number analyzed (Participants) | 0 | 21
  ALT, Day 1 | 0 | 0
  AST, Day 6: number analyzed (Participants) | 22 | 0
  AST, Day 6 | 0 | 0
  Cholesterol, Day 1 | 0 | 1
  Cholesterol, Day 6 | 1 | 1
  CRP, Day 1 | 0 | 0
  CRP, Day 6 | 1 | 0
  Hemoglobin decrease, Day 1 | 0 | 0
  Hemoglobin decrease, Day 6 | 0 | 0
  Haemoglobin, Day 1 | 0 | 0
  Haemoglobin, Day 6 | 0 | 0
  LDH, Day 6: number analyzed (Participants) | 22 | 0
  LDH, Day 6 | 0 | 0
  Neutrophils, Day 6 | 0 | 0
  RBC, Day 1 | 0 | 0
  RBC, Day 6 | 0 | 0
  Reticulocytes, Day 6: number analyzed (Participants) | 22 | 0
  Reticulocytes, Day 6 | 0 | 0
  WBC, Day 1 | 0 | 0
  WBC, Day 6: number analyzed (Participants) | 22 | 0
  WBC, Day 6 | 0 | 0
  Overall parameters, Day 1 | 0 | 1
  Overall parameters, Day 6 | 1 | 1

6. Secondary Outcome: Antibody Concentrations Against Pneumococcal Pneumolysin Toxoid (dPly) and Histidine Triad Protein D (PhtD) Proteins
Description: Anti-dPly and anti-PhtD antibody concentrations are presented as geometric mean concentrations (GMCs), expressed in LU/mL. The reference seropositivity cut-off values were equal to or above (≥) 599 LU/mL for anti-dPly and ≥ 391 LU/mL for anti-PhtD.
Time Frame: Prior to the booster vaccination (Day 0) and one month post-booster vaccination (Day 30)
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom post results were available for at least one assay.
Measure: Geometric Mean (95% Confidence Interval); unit: LU/mL
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 20
LU/mL
  Anti-dPly, Day 0 | 41823.0 [30264.0 to 57796.7] | 89612.2 [65851.0 to 121947.2]
  Anti-dPly, Day 30 | 92943.4 [65790.6 to 131302.6] | 144767.0 [106911.5 to 196026.4]
  Anti-PhtD, Day 0 | 26672.0 [19423.7 to 36625.0] | 42111.0 [33408.2 to 53080.9]
  Anti-PhtD, Day 30 | 37850.5 [29018.1 to 49371.2] | 62795.3 [51695.6 to 76278.3]

7. Secondary Outcome: Titers for Antibodies Against Pneumolysin Haemolysis (Hem-dPly) Protein
Description: Antibody titers are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 6.
Time Frame: Prior to the booster vaccination (Day 0) and one month post-booster vaccination (Day 30)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 20
Titers
  Anti-Hem-dPly, Day 0 | 2161.5 [1772.1 to 2636.4] | 3028.1 [2210.5 to 4148.1]
  Anti-Hem-dPly, Day 30 | 2383.6 [1754.4 to 3238.3] | 3573.7 [2561.1 to 4986.5]

8. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Any Pain | 19 | 21
  Any Redness | 4 | 9
  Any Swelling | 2 | 8

9. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhoea and/or abdominal pain), headache, malaise, myalgia and fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7-day (Days 0-6) post-booster vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Any Fatigue | 4 | 13
  Any Gastrointestinal symptoms | 3 | 1
  Any Headache | 5 | 8
  Any Malaise | 2 | 3
  Any Myalgia | 3 | 3
  Any Fever | 1 | 0

10. Secondary Outcome: Number of Subjects With Any Unsolicited AEs
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-booster vaccination period
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants | 6 | 5

11. Secondary Outcome: Number of Subjects With Any SAEs
Description: as for outcome 4
Time Frame: During the entire study period (from Day 0 to Day 30)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants | 0 | 0

12. Secondary Outcome: Number of Subjects With Grade 1, Grade 2 and Grade 4 Haematological or Biochemical Abnormalities
Description: as for outcome 5
Time Frame: At 1 and 6 days post-booster vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
Number analyzed (Participants) | 22 | 21
Participants
  Grade 1 ALT, Day 1: number analyzed (Participants) | 0 | 21
  Grade 1 ALT, Day 1 | 0 | 1
  Grade 1 AST, Day 6: number analyzed (Participants) | 22 | 0
  Grade 1 AST, Day 6 | 1 | 0
  Grade 1 Cholesterol, Day 1 | 3 | 4
  Grade 1 Cholesterol, Day 6 | 2 | 4
  Grade 1 CRP, Day 1 | 3 | 3
  Grade 1 CRP, Day 6 | 2 | 5
  Grade 1 Hemoglobin decrease, Day 1 | 7 | 7
  Grade 1 Hemoglobin decrease, Day 6 | 10 | 11
  Grade 1 Haemoglobin, Day 1 | 1 | 1
  Grade 1 Haemoglobin, Day 6 | 2 | 2
  Grade 1 LDH, Day 6: number analyzed (Participants) | 22 | 0
  Grade 1 LDH, Day 6 | 1 | 0
  Grade 1 Neutrophils, Day 6 | 2 | 2
  Grade 1 RBC, Day 1 | 7 | 5
  Grade 1 RBC, Day 6 | 6 | 4
  Grade 1 Reticulocytes, Day 6: number analyzed (Participants) | 22 | 0
  Grade 1 Reticulocytes, Day 6 | 1 | 0
  Grade 1 WBC, Day 1 | 2 | 3
  Grade 1 WBC, Day 6: number analyzed (Participants) | 22 | 0
  Grade 1 WBC, Day 6 | 1 | 0
  Grade 1 Overall parameters, Day 1 | 14 | 14
  Grade 1 Overall parameters, Day 6 | 17 | 17
  Grade 2 ALT, Day 1: number analyzed (Participants) | 0 | 21
  Grade 2 ALT, Day 1 | 0 | 0
  Grade 2 AST, Day 6: number analyzed (Participants) | 22 | 0
  Grade 2 AST, Day 6 | 0 | 0
  Grade 2 Cholesterol, Day 1 | 1 | 2
  Grade 2 Cholesterol, Day 6 | 1 | 2
  Grade 2 CRP, Day 1 | 1 | 1
  Grade 2 CRP, Day 6 | 2 | 1
  Grade 2 Hemoglobin decrease, Day 1 | 0 | 0
  Grade 2 Hemoglobin decrease, Day 6 | 0 | 0
  Grade 2 Haemoglobin, Day 1 | 1 | 0
  Grade 2 Haemoglobin, Day 6 | 1 | 0
  Grade 2 LDH, Day 6: number analyzed (Participants) | 22 | 0
  Grade 2 LDH, Day 6 | 0 | 0
  Grade 2 Neutrophils, Day 6 | 0 | 0
  Grade 2 RBC, Day 1 | 0 | 0
  Grade 2 RBC, Day 6 | 0 | 0
  Grade 2 Reticulocytes, Day 6: number analyzed (Participants) | 22 | 0
  Grade 2 Reticulocytes, Day 6 | 0 | 0
  Grade 2 WBC, Day 1 | 0 | 0
  Grade 2 WBC, Day 6: number analyzed (Participants) | 22 | 0
  Grade 2 WBC, Day 6 | 0 | 0
  Grade 2 Overall parameters, Day 1 | 3 | 3
  Grade 2 Overall parameters, Day 6 | 3 | 3
  Grade 4 ALT, Day 1: number analyzed (Participants) | 0 | 21
  Grade 4 ALT, Day 1 | 0 | 0
  Grade 4 AST, Day 6: number analyzed (Participants) | 22 | 0
  Grade 4 AST, Day 6 | 0 | 0
  Grade 4 Cholesterol, Day 1 | 0 | 0
  Grade 4 Cholesterol, Day 6 | 0 | 0
  Grade 4 CRP, Day 1 | 0 | 0
  Grade 4 CRP, Day 6 | 0 | 0
  Grade 4 Hemoglobin decrease, Day 1 | 0 | 0
  Grade 4 Hemoglobin decrease, Day 6 | 0 | 0
  Grade 4 Haemoglobin, Day 1 | 0 | 0
  Grade 4 Haemoglobin, Day 6 | 0 | 0
  Grade 4 LDH, Day 6: number analyzed (Participants) | 22 | 0
  Grade 4 LDH, Day 6 | 0 | 0
  Grade 4 Neutrophils, Day 6 | 0 | 0
  Grade 4 RBC, Day 1 | 0 | 0
  Grade 4 RBC, Day 6 | 0 | 0
  Grade 4 Reticulocytes, Day 6: number analyzed (Participants) | 22 | 0
  Grade 4 Reticulocytes, Day 6 | 0 | 0
  Grade 4 WBC, Day 1 | 0 | 0
  Grade 4 WBC, Day 6: number analyzed (Participants) | 22 | 0
  Grade 4 WBC, Day 6 | 0 | 0
  Grade 4 Overall parameters, Day 1 | 0 | 0
  Grade 4 Overall parameters, Day 6 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) follow-up period post-booster vaccination; Unsolicited AEs: during the 31-day (Days 0-30) follow-up period post-booster vaccination; SAEs: during the entire study period (from Day 0 up to Day 30).
Arm/Group | GSK2189242A Formulation 1 Group | GSK2189242A Formulation 2 Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 21/22 | 21/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2189242A Formulation 1 Group (N=22) | GSK2189242A Formulation 2 Group (N=21)
Pain (General disorders) | 19 | 21
Redness (General disorders) | 4 | 9
Swelling (General disorders) | 2 | 8
Fatigue (General disorders) | 4 | 13
Gastrointestinal symptoms (General disorders) | 3 | 1
Headache (General disorders) | 5 | 8
Malaise (General disorders) | 2 | 3
Myalgia (General disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Headache (Nervous system disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.